CLINICAL TRIAL: NCT05670522
Title: Transcranial Direct Current Stimulation Versus Virtual Reality on Gait in Children With Spastic Diplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Collaborators: Shirley Ryan AbilityLab (Other); Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Radwan, Assistant lecturer, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tDCS verus VR
Record Dates: First submitted 2022-12-06; First posted 2023-01-04 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Palsy
Keywords: Transcranial direct current stimulation; virtual reality; gait intervention; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial direct current stimulation group (Experimental): Children assigned to the transcranial direct current stimulation group received active transcranial direct current at their primary motor cortex (Active dose 11, ser. No 13070350, Active Tek Inc., USA). Stimulation was conducted at an intensity of 1 mA for 20 min per session, 5 times/week for 2 successive weeks (total of 10 sessions). 1 mA was shown to be appropriate in children's investigations. The anode (+) was positioned on the midline sagittal plane of the skull, corresponding to the motor area of lower limbs, and the cathode (-) was positioned over the inion. In addition to their assigned intervention, the children received the standard-of-care gait training. During the two-week intervention phase, gait training was administered immediately after each intervention session. Training was delivered in one hour increments 5 times/week for those first two weeks, then 3 times/week for the next 10 weeks.
  Interventions: Device: Transcranial direct current stimulation
- Virtual reality group (Experimental): Children assigned to the virtual reality group received virtual balance training using Nintendo Wii and Wii Balance Board, with a custom training program developed from activities on the Wii Fit Plus game. Training was conducted for 30 minutes, 5 sessions/week for 2 successive weeks (total of 10 sessions). Two sessions with Wii Fit Plus were conducted before the treatment protocol to help the children familiarize with the VR setup. In addition to their assigned intervention, the children received the standard-of-care gait training. During the two-week intervention phase, gait training was administered immediately after each intervention session. Training was delivered in one hour increments 5 times/week for those first two weeks, then 3 times/week for the next 10 weeks.
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct-current stimulation (tDCS), over the motor cortex, is a potential therapy option for motor control deficits in children with CP. The application of tDCS involves positioning 2 rubber electrodes sheathed in saline-soaked pads onto the scalp, held in place by a rubber strap. Low-intensity, direct-current, of 1 to 2 mA, is delivered to cortical areas from the device.
  The standard-of-care gait training included various gait training and balance tasks as well as resistive exercises and passive stretching as necessary. Task-specific gait exercises included: walking in a closed indoor environment, walking in an open indoor environment, walking on various floor surfaces, and climbing stairs up and down without assistance. The children also performed dynamic balance exercises by walking on a balance board.
  Arms: Transcranial direct current stimulation group
Device: Virtual reality — Virtual reality rehabilitation is an emerging therapy for motor rehabilitation of children with CP. The therapy is provided through a computer-simulated environment where they interact with real-world-like objects and events through sight, sound, and touch. The Wii Remote was used as the interactive interface, and standard computer/television screens were used as the display hardware. Therefore, VR therapy was of the non-immersive type.
  The standard-of-care gait training included various gait training and balance tasks as well as resistive exercises and passive stretching as necessary. Task-specific gait exercises included: walking in a closed indoor environment, walking in an open indoor environment, walking on various floor surfaces, and climbing stairs up and down without assistance. The children also performed dynamic balance exercises by walking on a balance board.
  Arms: Virtual reality group

SUMMARY:
Spastic diplegia is the most frequent type of cerebral palsy (CP), and impaired gait is a common sequela of this condition. The investigators compared the effects of two novel research interventions transcranial direct current stimulation (tDCS) and virtual reality (VR) on gait impairments in children with spastic diplegia.

Currently, both tDCS and VR require further investigation to determine their clinical effectiveness for children with CP. Thus, the aim of this study was to compare the effects of tDCS and VR training on spatiotemporal and kinetic gait parameters in children with spastic diplegia, as a supplemental intervention to traditional physical therapy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is caused by early-stage brain injury, affecting 2 to 3 children in every 1000 live births. CP is divided into different subtypes depending on the dominant neurological signs: spastic, dyskinetic, or ataxic. Epilepsy and intellectual disability, as well as problems with speech, hearing, and vision, are all common complications [1]. spastic diplegic CP is one of the most common developmental disabilities throughout life, caused by large-scale changes in subcortical brain activity with a reduced activation of corticospinal and somatosensory circuits, which leads to diminished activation of the central nervous system during volitional activities.

Gait impairment is seen in 90% of children with spastic diplegic CP, stemming from this decreased cortical excitability and compounded by spasticity of the lower extremities, excessive muscular weakness, impaired joint mobility, and poor coordination and balance. Specifically, children with CP have reduced gait velocity, cadence, and stride length, among other affected spatiotemporal gait parameters. The International Classification of Functioning Disability and Health consider changes in the spatial and temporal characteristics of gait to be important predictors to poor function and community participation. Additionally, crouched gait, scissoring, and other atypical gait patterns are common in this population, further affecting the kinematic and kinetic characteristics of gait and leading to metabolically expensive locomotion, high fall risk, and long-term musculoskeletal injury. For children with spastic diplegic CP, the primary goal of rehabilitation is to facilitate mobility and appropriate walking patterns with or without external assistance. Improving spatiotemporal and kinetic characteristics of gait would improve gait function, increase gait efficiency, and reduce the risk of long-term disability. In turn, it would allow these children to participate in more activities of daily living, meaningful interactions with family and society, and environmental exploration, as well as to improve their physical development.

In the current study, the investigators considered two technology-driven strategies that could potentially target gait impairments and improve gait function in children with CP: virtual reality (VR) and transcranial direct current stimulation (tDCS). Both interventions have been studied for their therapeutic potential with mixed results, especially in children. Specifically, VR can simulate real-life activities while providing repetition, augmented sensory input and feedback, error reduction/augmentation to increase motivation during the rehabilitation process. As a training tool, VR provides visual perceptual stimulation resulting from dynamic changes in context, which may aid in the execution of regulated exercises while also requiring concentration and additional postural control. Neuroimaging studies suggest that VR can facilitate learning and recovery by stimulating cortical reorganization and neural plasticity. Previous research has utilized VR as a therapeutic tool for children to improve balance, walking speed, and/or distance, as well as to encourage physical activity. Additional VR therapies have been shown to enhance functional performance in activities including squatting, standing posture, and energy expenditure. With the commercialization of VR-related products like the Nintendo Wii, many virtual games are readily available for home use. These games are often designed to challenge and train balance, posture, and dynamic movements all of which are critical factors for gait. Thus, VR-based rehabilitation may offer a unique, accessible therapeutic approach to reduce gait impairments and improve dynamic function.

In contrast, tDCS is a neuromodulation technique focused on optimizing existing neural pathways to prolong and/or improve the functional gains achieved by rehabilitation. tDCS is applied through either anodal or cathodal stimulation, which corresponds to excitation or inhibition of the stimulated brain areas, respectively. Anodal stimulation enhances cortical excitability through depolarization, allowing for more spontaneous cell firing, while cathodal stimulation has an inhibitory effect through hyperpolarization. Functionally, this means application of tDCS will influence activity in the area of the brain it targets. Previous research indicates that inhibited cortical input to the corticospinal tract is a possible cause of increased spasticity in CP, so it is reasonable to predict that anodal stimulation would mitigate these symptoms in individuals with spastic CP. The neurophysiological effects of anodal tDCS can also potentiate motor learning through this increase in cortical activity, which is applicable to the treatment of all subtypes of CP. These benefits may translate into functionally improved gait as well.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with diplegic CP
* the ages 7-12 years old
* minimum spasticity grades of 1 and 1+ according to modified Ashworth Scale
* Gross motor function classification system (GMFCS) at level I or II.
* Independent ambulation without any assistance or with minimal assistance
* A degree of cognition that allows understanding of the proposed procedures

Exclusion Criteria:

* children who had visual impairments, hearing damage, fixed deformities at lower limbs,
* History of orthopedic surgeries or injection with botulinum toxin in the previous year
* Had metal implants in the skull
* History of epilepsy or other neurological disorders
* or inability to understand the task.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-08-14 (Actual); Study Completion 2021-08-14 (Actual)

PRIMARY OUTCOMES:
Gait velocity (m/s) (Pre-treatment) | baseline
  Gait velocity was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with the soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Gait velocity (m/s) (post-treatment) | 2 weeks
  Gait velocity was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with the soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Gait velocity (m/s) (Follow up) | 10 weeks
  Gait velocity was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with the soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.

SECONDARY OUTCOMES:
Cadence (steps/min) (Pre-treatment) | Baseline
  Cadence was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Cadence (steps/min) (post-treatment) | 2 weeks
  Cadence was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Cadence (steps/min) (Follow up) | 10 weeks
  Cadence was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Stance time (s) (Pre-treatment) | Baseline
  Stance time was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Stance time (s) (post-treatment) | 2 weeks
  Stance time was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Stance time (s) (Follow up) | 10 weeks
  Stance time was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Swing time (s) (Pre-treatment) | Baseline
  Swing time was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Swing time (s) (post-treatment) | 2 weeks
  Swing time was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Swing time (s) (Follow up) | 10 weeks
  Swing time was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Step length (cm) (Pre-treatment) | Baseline
  Step length was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Step length (cm) (post-treatment) | 2 weeks
  Step length was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Step length (cm) (Follow up) | 10 weeks
  Step length was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Stride length (cm) (Pre-treatment) | Baseline
  Stride length was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Stride length (cm) (post-treatment) | 2 weeks
  Stride length was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Stride length (cm) (Follow up) | 10 weeks
  Stride length was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Maximum force (kg) (Pre-treatment) | Baseline
  Maximum force was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Maximum force (kg) (post-treatment) | 2 weeks
  Maximum force was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Maximum force (kg) (Follow up) | 10 weeks
  Maximum force was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Maximum peak pressure (N/cm²) (Pre-treatment) | Baseline
  Maximum peak pressure was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with the soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Maximum peak pressure (N/cm²) (post-treatment) | 2 weeks
  Maximum peak pressure was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.
Maximum peak pressure (N/cm²) (Follow up) | 10 weeks
  Maximum peak pressure was measured using Walkway Pressure Measurement System. This system consists of a digital mat inserted in a wooden walkway, equipped with sensors and a pressure recording system at a sampling resolution up to 185 Hz. A computer with soft-ware (version 7) and transmission hardware were used to download the data. Three trials were then completed to collect the gait parameters for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Hoda Eltalawy, PT, PhD, Principal Investigator — Cairo University, Egypt; Asmaa Radwan, PT, MSc, Principal Investigator — Beni-Suef University
Locations (1):
- outpatient clinic run by the faculty of physical therapy at Cairo University, Giza, Egypt

REFERENCES:
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598
- [Background] Hamilton A, Wakely L, Marquez J. Transcranial Direct-Current Stimulation on Motor Function in Pediatric Cerebral Palsy: A Systematic Review. Pediatr Phys Ther. 2018 Oct;30(4):291-301. doi: 10.1097/PEP.0000000000000535. PMID 30199513
- [Background] Saleem GT, Crasta JE, Slomine BS, Cantarero GL, Suskauer SJ. Transcranial Direct Current Stimulation in Pediatric Motor Disorders: A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2019 Apr;100(4):724-738. doi: 10.1016/j.apmr.2018.10.011. Epub 2018 Nov 7. PMID 30414398
- [Background] Grecco LA, Duarte NA, Zanon N, Galli M, Fregni F, Oliveira CS. Effect of a single session of transcranial direct-current stimulation on balance and spatiotemporal gait variables in children with cerebral palsy: A randomized sham-controlled study. Braz J Phys Ther. 2014 Sep-Oct;18(5):419-27. doi: 10.1590/bjpt-rbf.2014.0053. Epub 2014 Oct 10. PMID 25372004
- [Background] Ravi DK, Kumar N, Singhi P. Effectiveness of virtual reality rehabilitation for children and adolescents with cerebral palsy: an updated evidence-based systematic review. Physiotherapy. 2017 Sep;103(3):245-258. doi: 10.1016/j.physio.2016.08.004. Epub 2016 Sep 27. PMID 28109566
- [Background] Chen Y, Fanchiang HD, Howard A. Effectiveness of Virtual Reality in Children With Cerebral Palsy: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Phys Ther. 2018 Jan 1;98(1):63-77. doi: 10.1093/ptj/pzx107. PMID 29088476
- [Background] Warnier N, Lambregts S, Port IV. Effect of Virtual Reality Therapy on Balance and Walking in Children with Cerebral Palsy: A Systematic Review. Dev Neurorehabil. 2020 Nov;23(8):502-518. doi: 10.1080/17518423.2019.1683907. Epub 2019 Nov 1. PMID 31674852
- [Background] Biffi E, Beretta E, Storm FA, Corbetta C, Strazzer S, Pedrocchi A, Ambrosini E. The Effectiveness of Robot- vs. Virtual Reality-Based Gait Rehabilitation: A Propensity Score Matched Cohort. Life (Basel). 2021 Jun 11;11(6):548. doi: 10.3390/life11060548. PMID 34208009
- [Background] Valenzuela E, Rosa R, Monteiro C, Keniston L, Ayupe K, Fronio J, Chagas P. Intensive Training with Virtual Reality on Mobility in Adolescents with Cerebral Palsy-Single Subject Design. Int J Environ Res Public Health. 2021 Oct 5;18(19):10455. doi: 10.3390/ijerph181910455. PMID 34639757
- [Background] Kim CJ, Son SM. Comparison of Spatiotemporal Gait Parameters between Children with Normal Development and Children with Diplegic Cerebral Palsy. J Phys Ther Sci. 2014 Sep;26(9):1317-9. doi: 10.1589/jpts.26.1317. Epub 2014 Sep 17. PMID 25276007
- [Background] Corsi C, Santos MM, Moreira RFC, Dos Santos AN, de Campos AC, Galli M, Rocha NACF. Effect of physical therapy interventions on spatiotemporal gait parameters in children with cerebral palsy: a systematic review. Disabil Rehabil. 2021 Jun;43(11):1507-1516. doi: 10.1080/09638288.2019.1671500. Epub 2019 Oct 7. PMID 31588810